CLINICAL TRIAL: NCT01550549
Title: Evaluation of Web-based Training to Educate Physicians in the Methods of Interpreting Florbetapir-PET Scans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18F-AV-45-PT01
Record Dates: First submitted 2012-03-06; First posted 2012-03-12 (Estimated); Results first posted 2012-06-07 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-05

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Neurodegenerative Diseases
Keywords: Amyloid imaging; Positron Emission Tomography; 18F-AV-45; florbetapir F 18; Diagnostic imaging
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Neurodegenerative Diseases | interventions — florbetapir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: florbetapir F 18 — No study drug will be administered in this study - scans previously acquired in in Study A05(NCT00702143) and A07(NCT00857415) will be read
  Other Names: 18F-AV-45; Amyvid; florbetapir

SUMMARY:
This study will investigate the performance of physician readers trained to read florbetapir-PET scans using electronic media training.

DETAILED DESCRIPTION:
Avid has previously developed a florbetapir-PET scan binary read methodology and training program, which was successfully applied in studies 18F-AV-45-A08(NCT01565369), 18F-AV-45-A09(NCT01565382) and 18F-AV-45-A16(NCT01447719). In these previous studies, training was conducted in-person. Study 18F-AV-45-PT01 will evaluate an automated version of this training program suitable for web-based distribution. Nuclear medicine physicians will complete the automated training program then read the florbetapir-PET images from 151 subjects with repeat readings of 33 randomly selected images. Readers will rate each case as either positive for significant tracer accumulation in cortical gray matter or negative for significant tracer accumulation in cortical gray matter. The inter-rater reliability, sensitivity and specificity of the readers will be evaluated.

The primary image set for determination of inter-reader agreement is comprised of images from 119 subjects from two previous clinical studies (A07[NCT00857415]/A16[NCT01447719] and A05[NCT00702143]). This included all 59 subjects who came to autopsy in Study A07(NCT00857415) and it's follow-up study, A16(NCT01447719), and a set of 60 cases randomly selected from Study A05(NCT00702143) subjects, including 20 cognitively-normal controls, 20 with mild cognitive impairment) MCI, 20 with AD.

Subsequently, the protocol was amended to include all remaining A05(NCT00702143) MCI patients that were not used in the training program (n=32); 13 of these 32 scans presented for repeat reading (to increase the number of A05 MCI cases with repeated reads to 20). This increased the number of unique cases in the validation dataset to 151 scans with 33 scans repeated yielding a total of 184 scans reviewed by the readers.

ELIGIBILITY:
Eligibility for subjects scans to be used in this study is determined by subject's eligibility/enrollment in Study A05 (NCT00702143) or A07 (NCT00857415).

Alzheimer's disease (AD) group key eligibility criteria (from Study A05[NCT00702143]):

* Male or female at least 50 years of age
* Have probable AD per National Institute of Neurological and Communication Disorders and Stroke (NINCDS) criteria
* Mini mental state exam (MMSE) score between 10 and 24 inclusive

Mild cognitive impairment group key eligibility criteria (from Study A05[NCT00702143):

* Male or female at least 50 years of age
* Complaints of memory or cognitive decline corroborated by an informant
* Clinical dementia rating of 0.5
* No obvious cause for cognitive impairment (eg, head trauma or stroke)
* Cognitive impairment onset within the past year
* MMSE score greater than 24

Cognitively normal volunteer group key eligibility criteria (from Study A05[NCT00702143]):

* Male or female at least 50 years of age
* MMSE score greater than or equal to 29 and cognitively normal by informant report and psychometric test battery at screening

Autopsy cohort key eligibility criteria (from Study A07[NCT00857415]):

* Male or female 18 years or older
* Projected life expectancy of less than 6 months
* Consent to brain donation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals

RESULTS

PARTICIPANT FLOW:
Recruitment Details: NO SUBJECTS WERE ENROLLED IN THIS STUDY - this study re-read scans obtained in other clinical studies
Groups:
- Florbetapir-PET Scans: All subject scans with a valid florbetapir-PET scan
Period: Overall Study
Arm/Group | Florbetapir-PET Scans
Started | 151
Completed | 151
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Florbetapir-PET Scans: All subjects with a valid florbetapir-PET scan (59 from study A07/A16 and 92 from study A05)
Arm/Group | Florbetapir-PET Scans
Number analyzed (Participants) | 151
Age Continuous [Mean (Standard Deviation); unit: years] | 74.9 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75
  Male | 76
Region of Enrollment [Number; unit: participants]
  United States | 151

OUTCOME MEASURES:

1. Primary Outcome: Inter-rater Reliability
Description: Measure of agreement among five readers using a binary read method (amyloid positive/negative) calculated using Fleiss' kappa. All scans were read in a blinded fashion without access to clinical information.
Time Frame: Scan acquired 50-60 min post-injection
Population: 59 autopsy subjects (study A07[NCT00857415]/A16[NCT01447719]) + 20 healthy controls + 20 mild cognitive impairment + 20 AD (from study A05[NCT00702143])
Measure: Number (95% Confidence Interval); unit: kappa statistic
Arm/Group | Florbetapir-PET Scans Primary Analysis Group
Number analyzed (Participants) | 119
kappa statistic | 0.81 [0.75 to 0.87]

2. Secondary Outcome: Sensitivity of Florbetapir-PET to Detect Moderate to Frequent Beta-amyloid Neuritic Plaques (Probable/Definite Alzheimer's Disease)
Description: Calculated as the percent of true positives which are correctly identified
Time Frame: at autopsy, within 2 years of scan
Measure: Number (95% Confidence Interval); unit: percentage of positive cases IDed
Groups:
- All Autopsy: Subjects with a valid florbetapir-PET scan and autopsy (including those who deceased more than 12 months after the scan)
- Autopsy Within One Year of Scan: Subjects with a valid florbetapir-PET scan and autopsy (only those who deceased less than 12 months after the scan)
Arm/Group | All Autopsy | Autopsy Within One Year of Scan
Number analyzed (Participants) | 59 | 46
percentage of positive cases IDed
  Reader 1 | 79 [64.5 to 89.2] | 86 [68.5 to 94.3]
  Reader 2 | 92 [79.7 to 97.3] | 100 [87.9 to 100]
  Reader 3 | 69 [53.6 to 81.4] | 75 [56.6 to 87.3]
  Reader 4 | 87 [73.3 to 94.4] | 93 [77.4 to 98.0]
  Reader 5 | 82 [67.3 to 91.0] | 89 [72.8 to 96.3]

3. Secondary Outcome: Specificity of Florbetapir-PET to Detect no or Sparse Beta-amyloid Neuritic Plaques (Probable/Definite Alzheimer's Disease)
Description: Calculated as the percent of true negatives which are correctly identified
Time Frame: at autopsy, within 2 years of scan
Measure: Number (95% Confidence Interval); unit: percentage of negative cases IDed
Arm/Group | All Autopsy | Autopsy Within One Year of Scan
Number analyzed (Participants) | 59 | 46
percentage of negative cases IDed
  Reader 1 | 90 [69.9 to 97.2] | 89 [67.2 to 96.9]
  Reader 2 | 90 [69.9 to 97.2] | 89 [67.2 to 96.9]
  Reader 3 | 95 [76.4 to 99.1] | 94 [74.2 to 99.0]
  Reader 4 | 95 [76.4 to 99.1] | 94 [74.2 to 99.0]
  Reader 5 | 95 [76.4 to 99.1] | 100 [82.4 to 100]

4. Post Hoc Outcome: Inter-reader Reliability
Description: Measure of agreement among multiple readers using binary read method (Fleiss' kappa). Where available, histopathology analysis at autopsy was the truth standard (TS).
Time Frame: Scan acquired 50-60 min post-injection
Population: 59 from study A07(NCT00857415)/A16(NCT01447719) and 92 from study A05(NCT00702143)
Measure: Number (95% Confidence Interval); unit: kappa statistic
Groups:
- All Florbetapir-PET Scans: All subjects with a valid florbetapir-PET scan
Arm/Group | All Florbetapir-PET Scans
Number analyzed (Participants) | 151
kappa statistic
  All subjects [n=151] | 0.83 [0.78 to 0.88]
  All subjects with a TS [n=59] | 0.75 [0.67 to 0.83]
  All subjects without a TS [n=92] | 0.88 [0.82 to 0.94]
  AD [n=49] (29 with TS; 20 no TS) | 0.67 [0.58 to 0.76]
  MCI [n=57] (5 with TS; 52 no TS) | 0.91 [0.83 to 0.99]
  Cognitively normal without TS [n=20] | 0.83 [0.69 to 0.97]
  Cognitively normal with TS [n=12] | 0.73 [0.55 to 0.87]
  Other (non-AD) dementia with TS [n=13] | 0.52 [0.35 to 0.69]

5. Other Pre Specified Outcome: Median Sensitivity and Specificity vs. CERAD Diagnosis
Description: Median sensitivity and specificity for 5 independent readers to detect moderate to frequent amyloid plaques (per CERAD criteria).
Time Frame: Baseline scan
Measure: Median (Full Range); unit: percentage of true positives/negatives
Arm/Group | All Autopsy Population
Number analyzed (Participants) | 59
percentage of true positives/negatives
  Sensitivity | 82 [69 to 92]
  Specificity | 95 [90 to 95]

6. Post Hoc Outcome: Individual Reader Results (All Scans With Autopsy)
Description: Reader results (number of false negatives and number of false positives) for blinded independent readers. There were a total of 39 positive and 20 negative scans based on histopathology at autopsy.
Time Frame: Baseline scan
Measure: Number; unit: florbetapir scans
Groups:
- All Autopsy Population: Group of subjects with valid images who came to autopsy within 2 year of scan
Arm/Group | All Autopsy Population
Number analyzed (Participants) | 59
florbetapir scans
  Reader 1 - False Negatives | 8
  Reader 1 - False Positives | 2
  Reader 2 - False Negatives | 3
  Reader 2 - False Positives | 2
  Reader 3 - False Negatives | 12
  Reader 3 - False Positives | 1
  Reader 4 - False Negatives | 5
  Reader 4 - False Positives | 1
  Reader 5 - False Negatives | 7
  Reader 5 - False Positives | 1

7. Post Hoc Outcome: Individual Reader Results (Autopsy Within 1 Year of Scan)
Description: Reader results (number of false negatives and number of false positives) for blinded independent readers. There were a total of 28 positive and 18 negative scans based on histopathology at autopsy.
Time Frame: Baseline scan
Measure: Number; unit: florbetapir scans
Groups:
- Autopsy Within One Year of Scan: Group of subjects with valid images who came to autopsy within 1 year of scan
Arm/Group | Autopsy Within One Year of Scan
Number analyzed (Participants) | 46
florbetapir scans
  Reader 1 - False Negatives | 4
  Reader 1 - False Positives | 2
  Reader 2 - False Negatives | 0
  Reader 2 - False Positives | 2
  Reader 3 - False Negatives | 7
  Reader 3 - False Positives | 1
  Reader 4 - False Negatives | 2
  Reader 4 - False Positives | 1
  Reader 5 - False Negatives | 3
  Reader 5 - False Positives | 0

ADVERSE EVENTS:
Description: No subjects received florbetapir in this study. This study consisted of re-reads of scans previously acquired in other clinical studies (A05, A07, A16).
Arm/Group | Florbetapir-PET Scans
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days